CLINICAL TRIAL: NCT01878786
Title: A Pilot Study Comparing the Safety and Efficacy of Zortress (Everolimus) With Low Dose Tacrolimus to Early Conversion to Calcineulin Inhibitor-Free Regimen and Mycophenolic Acid With Standard Dose Tacrolimus in Recipients of ECD/DCD Kidneys
Brief Title: A Pilot Study Comparing the Safety and Efficacy of Everolimus With Other Medicines in Recipients of ECD/DCD Kidneys
Acronym: Evered
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Interim results suggested a concern for patient outcomes and safety
Sponsor: Matthew Cooper (Other)
Responsible Party: Sponsor-Investigator, Matthew Cooper, Dr. Matthew Cooper, Georgetown University
Organization: Georgetown University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIRPCRAD001AUS183T
Record Dates: First submitted 2013-06-11; First posted 2013-06-17 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Delayed Graft Function
Keywords: kidney failure
MeSH Terms: conditions — Delayed Graft Function; Renal Insufficiency | interventions — Everolimus; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ERL & TAC (Experimental): Concentration controlled everolimus(ERL) & Low dose tacrolimus(TAC) + corticosteroid withdraw
  Interventions: Drug: Everolimus; Drug: Tacrolimus
- ERL & TAC --> MMF/MPA (Experimental): Concentration controlled everolimus & low dose tacrolimus --> mycophenolate mofetil (MMF) at Month 3 + corticosteroid
  Interventions: Drug: Everolimus; Drug: Tacrolimus; Drug: Mycophenolate mofetil (MMF/MPA)
- Standard dose TAC + MMF/MPA (Experimental): Standard dose of tacrolimus + mycophenolate mofetil + corticosteroid withdraw
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate mofetil (MMF/MPA)

INTERVENTIONS:
Drug: Everolimus — One of the immunosuppressants currently being evaluated to replace CNIs in patients with CNI nephropathy is the mammalian Target of Rapamycin (mTOR) inhibitor, Sirolimus. Everolimus is a derivative of Sirolimus and belongs to this class of immunosuppressants, therefore, both drugs have similar side effect profile. The half-life of Everolimus is almost half of Sirolimus (Everolimus 30 hours vs Sirolimus 62 hours), which makes its dose adjustment easier although it would require more frequent dosing. In clinical trials, Everolimus has demonstrated its potential role as a safe alternative in minimizing and/or eliminating CNI such as Cyclosporin A and Tacrolimus .
  Other Names: Zortress
  Arms: ERL & TAC; ERL & TAC --> MMF/MPA
Drug: Tacrolimus — One of the immunosuppressants currently being evaluated to replace CNIs in patients with CNI nephropathy is the mammalian Target of Rapamycin (mTOR) inhibitor, Sirolimus. Everolimus is a derivative of Sirolimus and belongs to this class of immunosuppressants, therefore, both drugs have similar side effect profile. The half-life of Everolimus is almost half of Sirolimus (Everolimus 30 hours vs Sirolimus 62 hours), which makes its dose adjustment easier although it would require more frequent dosing. In clinical trials, Everolimus has demonstrated its potential role as a safe alternative in minimizing and/or eliminating CNI such as Cyclosporin A and Tacrolimus.
  Other Names: Prograf
Drug: Mycophenolate mofetil (MMF/MPA) — Control Drug
  Other Names: CellCept
  Arms: ERL & TAC --> MMF/MPA; Standard dose TAC + MMF/MPA

SUMMARY:
The purpose of this pilot study is to evaluate concentration-controlled everolimus with low dose tacrolimus compared to early conversion to CNI-free regimen and MMF/MPA with standard dose tacrolimus in de novo renal transplant recipients of ECD/DCD kidneys. Given tacrolimus and MMF/MPA is a widely prescribed immunosuppressive regimen in the United States, comparisons of tacrolimus and MMF/MPA regimens to investigational therapies and treatment regimens are needed. Also, considering the fact that ECD/DCD is a fast growing fraction of donors, evaluation of various regimens' effects on rather delicate ECD/DCD kidneys is necessary.

DETAILED DESCRIPTION:
The purpose of this pilot study is to evaluate concentration-controlled everolimus with low dose tacrolimus compared to early conversion to CNI-free regimen and MMF/MPA with standard dose tacrolimus in de novo renal transplant recipients of ECD/DCD kidneys. Given tacrolimus and MMF/MPA is a widely prescribed immunosuppressive regimen in the United States, comparisons of tacrolimus and MMF/MPA regimens to investigational therapies and treatment regimens are needed. Also, considering the fact that ECD/DCD is a fast growing fraction of donors, evaluation of various regimens' effects on rather delicate ECD/DCD kidneys is necessary.

The primary objective of this study is to evaluate concentration-controlled everolimus and low dose tacrolimus compared to MMF/MPA with standard dose tacrolimus at 24 months post-transplant with respect to the composite efficacy failure rates (treated biopsy proven acute rejection episodes (BPAR), graft loss, death, loss to follow-up) in de novo renal transplant recipients.

The key secondary objective is to compare renal function of the everolimus treatment arms to the MMF/MPA treatment arm at 12 and 24 months post-transplantation. Renal function will be measured by the calculated glomerular filtration rate (GFR), using the MDRD (Modification of Diet in Renal Disease) formula (20).

ELIGIBILITY:
Inclusion Criteria:

Male or female recipients 18-65 years of age undergoing primary or secondary kidney transplantation

Recipients of primary or secondary cadaveric, ECD/DCD kidney (defined as follows)

Donor whose heart has irreversibly stopped beating, previously referred to as non-heart-beating or asystolic donation

Brain-dead donor > 60 years old

Donor aged 50-59 years old with two of the following criteria:

History of hypertension

Terminal serum creatinine ≥ 1.5 mg/dL

Death resulting from cerebrovascular accident

Patients who have given written informed consent to participate in the study

Exclusion Criteria:

Cold ischemic time (CIT) > 30 hours

Patients who are ABO incompatible transplants, or T, or B cell crossmatch positive transplant

Patients with a known hypersensitivity to any of the study drugs or to drugs of similar chemical class

Non-controlled DCD

Donor age >70

Patients with BMI >32 at baseline before surgery

Pregnant or lactating females

Females of childbearing potential unwilling to use an effective means of contraception or are planning to become pregnant

Patients with platelet count <100,000/mm3 at the evaluation before randomization.

Patients with an absolute neutrophil count of < 1,500/mm³ at baseline before surgery or white blood cell count of < 4,500/mm³

Patients who are recipients of multiple solid organ transplants

Patients who have severe hypercholesterolemia (>350 mg/dL; >9 mmol/L) or hypertriglyceridemia (>500 mg/dL; >5.6 mmol/L). Patients with controlled hyperlipidemia are acceptable

Patients who have an abnormal liver profile such as ALT, AST, Alk Phos or total bilirubin >3 times the upper normal limit

Patients who are treated with drugs that are strong inducers or inhibitors of cytochrome P450 3A4, such as terfenadine, astemizole, cisapride, erythromycin, azithromycin, itraconazole, rifampin or lovastatin

Patients who received an investigational drug or who have been treated with a non-protocol immunosuppressive drug or treatment within 30 days or 5 half-lives prior to randomization

Patients with a history of malignancy of any organ system, treated or untreated, within the past 2 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin

Patients who are HIV-positive or Hepatitis C (PCR+ only) or B surface antigen positive

Recipients of organs from donors who test positive for Hepatitis B surface antigen or Hepatitis C (PCR+ only) are excluded

Patients with a history of severe diarrhea, active peptic ulcer disease, or uncontrolled diabetes mellitus (Hgb A1c <7.0 %) at baseline

Patients who have any surgical or medical condition, which in the opinion of the investigator, might significantly alter the absorption, distribution, metabolism and excretion of study medication, and/or the presence of severe diarrhea or active peptic ulcer

Patients who have cardiac failure (e.g. resting dyspnea, symptoms with less than ordinary activity, marked limitation of activity) at time of screening or any other severe cardiac disease as determined by the investigator

Patients with abnormal physical or laboratory findings of clinical significance within 3 months of randomization which would interfere with the objectives of the study

Patients with any history of coagulopathy or medical condition requiring long-term anticoagulation therapy after transplantation (Low dose aspirin treatment is allowed)

Patients with known history of focal segmental glomeruloscrelosis

Presence of psychiatric illness (i.e., schizophrenia, bipolar, major depression) that, in the opinion of the investigator, would interfere with study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-06; Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Cooper, Principal Investigator — Georgetown University Hospital
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ERL & TAC: Concentration controlled everolimus(ERL) & Low dose tacrolimus(TAC) + corticosteroid withdraw
  Everolimus: One of the immunosuppressants currently being evaluated to replace CNIs in patients with CNI nephropathy is the mammalian Target of Rapamycin (mTOR) inhibitor, Sirolimus. Everolimus is a derivative of Sirolimus and belongs to this class of immunosuppressants, therefore, both drugs have similar side effect profile. The half-life of Everolimus is almost half of Sirolimus (Everolimus 30 hours vs Sirolimus 62 hours), which makes its dose adjustment easier although it would require more frequent dosing. In clinical trials, Everolimus has demonstrated its potential role as a safe alternative in minimizing and/or eliminating CNI such as Cyclosporin A and Tacrolimus .
  Tacrolimus: CNI
- ERL & TAC --> MMF/MPA: Concentration controlled everolimus & low dose tacrolimus --> mycophenolate mofetil (MMF) at Month 3 + corticosteroid withdraw
  Everolimus: One of the immunosuppressants currently being evaluated to replace CNIs in patients with CNI nephropathy is the mammalian Target of Rapamycin (mTOR) inhibitor, Sirolimus. Everolimus is a derivative of Sirolimus and belongs to this class of immunosuppressants, therefore, both drugs have similar side effect profile. The half-life of Everolimus is almost half of Sirolimus (Everolimus 30 hours vs Sirolimus 62 hours), which makes its dose adjustment easier although it would require more frequent dosing. In clinical trials, Everolimus has demonstrated its potential role as a safe alternative in minimizing and/or eliminating CNI such as Cyclosporin A and Tacrolimus .
  Tacrolimus: One of the immunosuppressants currently being evaluated to replace CNIs in patients with CNI nephropathy is the mammalian Target of Rapamycin (mTOR) inhibitor, Sirolimus.
Period: Overall Study
Arm/Group | ERL & TAC | ERL & TAC --> MMF/MPA | Standard Dose TAC + MMF/MPA
Started | 9 | 9 | 7
Completed | 0 (Study closed prematurely) | 0 (Study closed prematurely) | 0 (Study closed prematurely; 1 patient was a screen fail)
Not Completed | 9 | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ERL & TAC | ERL & TAC --> MMF/MPA | Standard Dose TAC + MMF/MPA | Total
Number analyzed (Participants) | 9 | 9 | 7 | 25
Age, Categorical [Count of Participants; unit: Participants] — Population: 24 patients were between 18 and 65, one patient 65
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 9 | 9 | 6 | 24
    >=65 years | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 8
  Male | 6 | 6 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 8 | 8 | 7 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 6 | 7 | 21
  White | 0 | 2 | 0 | 2
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Concentration-controlled Everolimus and Low Dose Tacrolimus Compared to MMF/MPA With Standard Dose Tacrolimus at 24 Months
Description: The primary objective of this study is to evaluate concentration-controlled everolimus and low dose tacrolimus compared to MMF/MPA with standard dose tacrolimus at 24 months post-transplant with respect to the composite efficacy failure rates (treated biopsy proven acute rejection episodes (BPAR), graft loss, death, loss to follow-up) in de novo renal transplant recipients.
Time Frame: 24 months
Population: Study was terminated prematurely. There was no data analysis performed on the incomplete data set.
Arm/Group | ERL & TAC | ERL & TAC --> MMF/MPA | Standard Dose TAC + MMF/MPA
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Compare Renal Function of the Everolimus Treatment Arms to the MMF/MPA Treatment Arm at 12 and 24 Months Post-transplantation
Description: The key secondary objective is to compare renal function of the everolimus treatment arms to the MMF/MPA treatment arm at 12 and 24 months post-transplantation. Renal function will be measured by the calculated glomerular filtration rate (GFR), using the MDRD (Modification of Diet in Renal Disease) formula (20).
Time Frame: 24 months
Population: Study was terminated prematurely. There was no data analysis performed on the incomplete data set.
Arm/Group | ERL & TAC | ERL & TAC --> MMF/MPA | Standard Dose TAC + MMF/MPA
Number analyzed (Participants) | 0 | 0 | 0

3. Other Pre Specified Outcome: Incidence of Cytomegalovirus (CMV) (Viremia or Viruria)
Time Frame: 24 months
Population: Study was terminated prematurely. There was no data analysis performed on the incomplete data set.
Arm/Group | ERL & TAC | ERL & TAC --> MMF/MPA | Standard Dose TAC + MMF/MPA
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of study drug through the end of the study. The study was terminated prematurely.
Arm/Group | ERL & TAC | ERL & TAC --> MMF/MPA | Standard Dose TAC + MMF/MPA
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 7/9 | 2/9 | 2/7
Other Adverse Events (participants affected / at risk) | 8/9 | 9/9 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ERL & TAC (N=9) | ERL & TAC --> MMF/MPA (N=9) | Standard Dose TAC + MMF/MPA (N=7)
Sepsis and Multiple Organ Failure (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GI Surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Left Renal Mass/Nephrectomy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Neck and Facial Edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Admission (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
ER Admission for Blood Transfusion (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
UTI (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Possible malrotation of kidney, possible uretropelvic junction obstruction) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Fluid Overload and Chest Pressure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wound Dehiscence (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ERL & TAC (N=9) | ERL & TAC --> MMF/MPA (N=9) | Standard Dose TAC + MMF/MPA (N=7)
Acute Rejection (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
CMV (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
BK Viuria (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
BK Viremia (Infections and infestations) | 3 (3) | 2 (2) | 2 (2)
Oral Candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Penile Edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Epididymo-Orchitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Scrotal Edema (General disorders) | 1 (1) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urothelial Papilloma (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Testicular Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (5) | 6 (6) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 5 (5)
CNI Toxicity (Investigations) | 1 (1) | 0 (0) | 0 (0)
Elevated Serum Creatinine (Investigations) | 1 (1) | 2 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Anasarca (General disorders) | 1 (1) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 3 (3) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Neck Edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Facial Edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Delayed Graft Function (Renal and urinary disorders) | 1 (1) | 4 (4) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Borderline ACR (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Wound Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Antibody Mediated Rejection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Poor Wound Healing (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Localized Edema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Acute Cellular Rejection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Itching Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Burning Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Worsening Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lower Extremity Edema (General disorders) | 0 (0) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Diaphoresis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
NODAT (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Submandibular Abscess (General disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Liver Injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Sickle Cell Crisis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely and analysis was not performed on the incomplete data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT01878786/Prot_SAP_000.pdf